CLINICAL TRIAL: NCT01627717
Title: The Effects of the Direct Acting Antiviral Agent Boceprevir on the Pharmacokinetics of Maraviroc in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: Université de Montréal (Other); McGill University Health Centre/Research Institute of the McGill University Health Centre (Other); Toronto General Hospital (Other)
Responsible Party: Principal Investigator, Nancy Sheehan, Associate Clinical Professor, Centre hospitalier de l'Université de Montréal (CHUM)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: MVC.1201
Record Dates: First submitted 2012-06-21; First posted 2012-06-26 (Estimated); Last update posted 2018-01-26 (Actual); Status verified 2018-01

CONDITIONS: Healthy
Keywords: maraviroc; boceprevir; HIV; HCV; drug interaction; pharmacokinetics
MeSH Terms: interventions — Maraviroc; N-(3-amino-1-(cyclobutylmethyl)-2,3-dioxopropyl)-3-(2-((((1,1-dimethylethyl)amino)carbonyl)amino)-3,3-dimethyl-1-oxobutyl)-6,6-dimethyl-3-azabicyclo(3.1.0)hexan-2-carboxamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Maraviroc Boceprevir (Experimental)
  Interventions: Drug: Maraviroc (5 days); Drug: Maraviroc and boceprevir (14 days)

INTERVENTIONS:
Drug: Maraviroc (5 days) — Subjects will receive maraviroc 150 mg tablets (1 tablet) every 12 hours from days 1 to 5 inclusively.
  Other Names: Celsentri (DIN #: 02299844) CAS# 376348-65-1
Drug: Maraviroc and boceprevir (14 days) — From days 6 to 19, inclusively, boceprevir 800 mg (4 capsules of 200 mg) every 8 hours with food will be given with maraviroc 150 mg (1 tablet of 150 mg) every 12 hours.
  Other Names: Celsentri (DIN #: 02299844) CAS# 376348-65-1; Victrelis (DIN#:02370816) CAS# 394730-60-0

SUMMARY:
Infection by both HIV and hepatitis C virus (HCV)is frequent due to similar transmission modes. Near 20% of people living with HIV are also infected by HCV. People living with HIV are treated by anti-HIV medications that may interact with numerous other medications, including new medications against HCV.

Boceprevir is one of these new HCV medications and it is now considered as part of the standard of care for people infected with HCV. Previous research has shown boceprevir may influence the capacity of the liver to breakdown (metabolize) certain medications and when these medications are used in combination with boceprevir, their blood concentrations may be increased or decreased which could increase the risk of side effects or decrease efficacy. Among the drugs having a potential for an interaction with boceprevir is maraviroc, an anti-HIV medication. If concentrations of maraviroc increase, people may experience more side effects. However, if concentrations of maraviroc decrease, people living with HIV may have a lower suppression of the virus. This could increase the risk for the HIV virus to develop resistance, that is that the treatment will no longer be effective. No studies have been conducted to investigate the effects of boceprevir on blood concentrations of maraviroc. This research project addresses this research question. This project, however, cannot be done with people living with HIV since resistance may develop in these people if the concentrations of maraviroc decrease. It is for this reason that the investigators wish to recruit healthy people not infected with HIV nor HCV.

Eleven healthy volunteers will be included. They will receive maraviroc 150 mg (1 tablet) every 12 hours from days 1 to 19 inclusively. On day 5, a total of ten blood samples will be drawn during the following 12 hours (at 0, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8 and 12 hours after maraviroc morning dose intake) to measure the blood concentrations of maraviroc. Boceprevir 800 mg (4 capsules) every 8 hours with food will be started on day 6 and continued until day 19 inclusively. On day 19, after the morning maraviroc and boceprevir dose, another ten blood samples will be drawn over a 12 hour period. A phone follow-up will be done on day 26. Thus, the total study duration for subjects is 26 days. The investigators will compare the blood concentrations of maraviroc when given alone to the blood concentrations of maraviroc when given with boceprevir.

DETAILED DESCRIPTION:
Co-infection with human immunodeficiency virus (HIV) and hepatitis C virus (HCV) is frequent because of shared modes of viral transmission. Near 20% of HIV-infected patients are also infected with HCV, the prevalence of HCV in the HIV population varying according to the route of transmission. Despite the decrease in mortality and morbidity in HIV-infected individuals since the introduction of potent combination antiretroviral therapy (cART), HCV-related end-stage liver disease (ESLD) now represents a leading cause of death in these patients.

HCV treatment outcomes in terms of sustained virologic response (SVR) are usually worse in co-infected patients, pegylated interferon-alpha (PEG IFN-alpha) / ribavirin treatment leading to success in only 40 to 50% of mono-infected patients and 30 % of co-infected patients. In patients co-infected with HIV, present guidelines recommend a fixed course of PEG IFN-alpha / ribavirin for 48 weeks to optimize HCV treatment.

The recent introduction of boceprevir and telaprevir, two direct acting antiviral agents (DAAs) against HCV, changed the standard of care for the treatment of chronic HCV infection with genotype 1, whereby now the AASLD practice guidelines recommend the use of boceprevir or telaprevir in combination with PEG IFN-alpha/ribavirin in both HCV mono-infected treatment naïve and experienced patients. No studies have yet been published in HCV-HIV co-infected patients.

Boceprevir is a novel HCV NS3 serine protease inhibitor (PI). In clinical studies of treatment-naïve and experienced patients, this agent, in combination with standard of care (PEG IFN-alpha/ribavirin), achieved much greater SVR rates, reaching rates higher than 70 % in clinical studies.

Boceprevir has to be taken 800 mg (four 200 mg capsules) three times a day (every 7-9 hours) with food. Boceprevir is usually well tolerated according to single and multiple dose pharmacokinetics studies in healthy volunteers with adverse effects similar to placebo. The serious adverse effects related to boceprevir are seen when boceprevir is coadministered with PEG-IFN alpha/ribavirin. These include anemia, neutropenia and thrombocytopenia.

An interim analysis of a randomized double-blind placebo-controlled study of the use of boceprevir/PEG IFN-alpha/ribavirin in HCV treatment naïve HCV/HIV co-infected patients showed that 70.5 % of patients on boceprevir/PEG IFN-alpha/ribavirin had an undetectable HCV RNA at 24 weeks as compared to 34.4% of patients on PEG IFN-alpha/ribavirin.

Boceprevir metabolism is mediated mainly by aldo-keto reductases and by CYP3A4 and CYP3A5. Boceprevir is also a substrate of p-glycoprotein (P-gp). Boceprevir is by itself known to be a strong inhibitor of CYP3A4/3A5 and drugs metabolized by this pathway may have increased exposure when administered with this product. In vitro data has shown that boceprevir does not induce CYP3A4/5. Surprisingly, however, a recent warning by the FDA (FDA Medwatch, February 9th 2012) and a Dear Health Care Professional Letter from Merck & Co, Inc. (USA) have revealed that boceprevir decreases the exposure of HIV ritonavir-boosted protease inhibitors that are CYP3A4 substrates. This unpublished data suggests that boceprevir in vivo may be acting as a CYP3A4 inducer. Contradictory in vitro and in vivo drug interaction study results are not uncommon. The clinical impact of these interactions is at the moment unclear. This has implications for possible drug-drug interactions if boceprevir is used in combination with cART in HIV/HCV co-infected patients.

Among the antiretroviral drugs that seem promising to be used in HIV/HCV co-infected patients is maraviroc. A recent conference abstract suggests that adding maraviroc to an antiretroviral regimen in HIV/HCV-co-infected patients naïve to anti-HCV therapy decreases liver fibrosis. Maraviroc is usually given as 300 mg twice daily with or without food but the dose may change depending on the patient's concomitant medications. Maraviroc does not inhibit any of the major CYP450 enzymes (CYP1A2, CYP2B6, CYP2C8, CYP2C9, CYP2C19, CYP2D6 and CYP3A4) and does not show any effects on plasma concentrations of other molecules. Maraviroc's major metabolic routes are oxidation and N-dealkylation and in vitro studies demonstrated that maraviroc is primarily metabolized by CYP3A4. Concomitant use of maraviroc with known CYP3A4 inhibitors requires maraviroc dosage to be reduced to 150 mg twice a day while its use with CYP3A4 inducers necessitates maraviroc to be used 600 mg twice daily.

Maraviroc was well tolerated in the various clinical trials with a drop-out rate of 4 to 6 % similar to placebo. The most common side effects are upper respiratory tract infections (22,8 %), cough (13,8%), fever (12,9 %), rash (10,8 %), muscle-related symptoms (9,9 %), dizziness and postural dizziness (8,7 %), abdominal pain (8.2 %), insomnia (7,7 %) and constipation (5,9%) (19). Maraviroc should be used with caution in patients with an increased risk of cardiovascular events as cases of myocardial infarction, postural hypotension and syncope have been reported. Postural hypotension is dose-related and unlikely to occur at labeled doses. However, postural hypotension may be of concern if drug-drug interactions occur without proper dose adjustments of maraviroc. The use of maraviroc 150 mg BID in steady-state drug-drug interaction studies in healthy volunteers in the presence of potent CYP3A4 inhibitors has been well tolerated.

No study regarding the use of maraviroc with boceprevir has been conducted. Given the similar metabolic routes taken by these molecules, that is CYP3A4, it is likely that these molecules will interact. It is unknown if boceprevir will increase or decrease maraviroc systemic exposure. To limit potential toxicity and study discontinuations, however, we have chosen to do the study with maraviroc 150 mg twice daily. The study will evaluate the effects of boceprevir on the pharmacokinetics of maraviroc in healthy volunteers. As maraviroc does not inhibit nor induce CYP 450 isoenzymes, maraviroc is not expected to influence boceprevir pharmacokinetics. For this reason, we have chosen not to measure boceprevir concentrations.

This is a phase 1, single center, open-label, crossover single-sequence drug-drug interaction study in healthy Caucasian males. The study population is limited to Caucasian males to limit interpatient pharmacokinetic variability. Eleven healthy volunteers will be included. They will receive maraviroc 150 mg every 12 hours from days 1 to 19 inclusively. On day 5, 12 hour intensive pharmacokinetic sampling will be done to measure maraviroc in the absence of boceprevir. Boceprevir 800 mg every 8 hours with food will be started on day 6 and continued until day 19 inclusively. On day 19, 12 hour intensive pharmacokinetic sampling will be repeated to measure maraviroc concentrations in the presence of boceprevir. The maraviroc concentration will be at steady-state by day 5. Furthermore, 14 days of boceprevir will be sufficient to study inhibition and induction. A phone follow-up will be done on day 26. Thus, the total study duration for subjects is 26 days.

The primary objective of the study is to evaluate the effects of boceprevir on the pharmacokinetics of maraviroc in healthy volunteers. The secondary objective is to determine the appropriate maraviroc dose to be taken when given concomitantly with boceprevir.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian males
* healthy individuals based on history/physical examination and laboratory evaluations (no out-of-range results from hematology tests (hemoglobin (Hb) > 130 g/L in men; absolute neutrophil count (ANC) > 2000 cells/uL; platelets > 159 x 109/L), biochemistry (AST < 35 IU/L, ALT < 40, IU/L, alkaline phosphatase < 100 IU/L, total bilirubin < 17 umol/L, lipase < 45 IU/L, creatinine < 120 umol/L, normal coagulation tests (INR < 1.2, aPPT < 40 seconds) and urinalysis.
* LDL-cholesterol </= 5 mmol/L, triglycerides </= 1.7 mmol/L and a 10 year estimate of cardiovascular (CV) disease risk of </= 10% ("low risk") as per the Framingham risk score modified for family history (doubling of CV risk if any CV disease in a first-degree relative before 60 years of age); the modified Framingham risk score takes into account age, HDL-cholesterol, total cholesterol, systolic blood pressure, smoker status, presence of diabetes and family history of CV disease
* normal 12-lead electrocardiogram
* systolic blood pressure between 105 and 130 mmHg
* diastolic blood pressure between 60 and 90 mmHg
* supine heart rate between 60 and 100 beats per minutes
* no evidence of HIV infection (ELISA test and Western Blot), no evidence of hepatitis B virus infection (HBsAg negative and anti-HBcAg negative or HBsAg negative with positive anti-HBsAg and positive anti-HBcAg) or HCV infection at screening (anti-HCV serology)
* using an effective barrier method of contraception
* non-smoker
* drinking less than 14 units of alcohol per week with a maximum of 4 units per day where one unit of alcohol corresponds to 341 mL of standard beer or 142 mL of wine or 43 ml of spirits
* negative illicit drug test at screening;
* with a body mass index between 18.0 to 30.0 kg/m2
* aged from 18 to 50 years old
* volunteers must be able to understand and comply with the protocol requirements and willing to sign the informed consent form prior to any study procedure;
* absence of exclusion criteria.

Exclusion Criteria:

* history of postural hypotension
* cardiac disease
* acute or chronic liver disease or any hepatic impairment
* acute or chronic kidney disease or any renal impairment
* use of prescription drugs, over the counter drugs, recreational drugs, herbal or dietary supplements including vitamins and grapefruit juice within 15 days of study initiation (day 1) except for acetaminophen and/or ibuprofen on an as needed basis. These products will also be prohibited during the study (except for as needed acetaminophen and/or ibuprofen)
* subjects who received any experimental medication within the last 2 months and/or donated blood during the previous 2 months or intends to donate blood within 2 months following completion of the study will also be excluded;
* subjects who had unprotected sexual activities during the last 6 months with a new or recent partner
* subjects who injected intravenous drugs over the last 6 months
* subjects with a social condition, psychological or addictive disorder that would impair protocol adherence.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2012-06; Primary Completion 2013-04 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Change in maraviroc AUC | Day 19

SECONDARY OUTCOMES:
Change in maraviroc Tmax | Day 19
Adverse events | Up to day 26
  Adverse events will be graded according to the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events (2004).
Change in maraviroc Cmax | Day 19
Change in maraviroc Cmin | Day 19
Change in maraviroc Cl/F | Day 19
Change in maraviroc Vd | Day 19
Change in maraviroc T1/2 | Day 19

CONTACTS AND LOCATIONS:
Overall Officials: Cecile Tremblay, MD, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM); Line Labbé, PhD, Principal Investigator — Faculté de pharmacie, Université de Montréal; Nancy L Sheehan, B.Pharm, MSc, Principal Investigator — Faculté de pharmacie, Université de Montréal; Alice Tseng, PharmD, Study Director — Toronto General Hospital
Locations (1):
- Centre Hospitalier de l'Université de Montréal, Montreal, Quebec, Canada